CLINICAL TRIAL: NCT00692575
Title: Modular Scheduled Telephone Intervention for Caregivers of Persons With Traumatic Brain Injury: A Randomized Controlled Trial
Brief Title: Telephone Intervention for Caregivers of Persons With Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janet Powell, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33690-J; NIDRR grant # H133A070032 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Brain Injuries
Keywords: Brain Injuries, Traumatic; Caregivers
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Experimental (Experimental): Problem-solving, education based telephone counseling.
  Interventions: Behavioral: Problem-solving, education based telephone counseling
- 2: No intervention (Sham Comparator): Standard of care control group
  Interventions: Other: No Intervention

INTERVENTIONS:
Behavioral: Problem-solving, education based telephone counseling — Caregivers are contacted every 2 weeks for 16-20 weeks after discharge of TBI survivor home. A caregiver support specialist provides telephone counseling based on a problem-solving, educational model.
  Arms: 1: Experimental
Other: No Intervention — The control group will receive standard of care, i.e., typical resources and/or supports offered to caregivers of persons with TBI.
  Other Names: Standard of care
  Arms: 2: No intervention

SUMMARY:
This study seeks to determine if problem-based telephone counseling improves quality of life and emotional well-being for caregivers of persons with moderate to severe traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Caregivers and patients with TBI are recruited from the acute medical and inpatient rehabilitation units at Harborview Medical Center and the University of Washington Medical Center in Seattle, WA. After informed consent is obtained, information is gathered from the caregiver about his/her living situation, support systems, and the nature of the caregiving relationship. Additional information is gathered from the person with TBI about how he/she is doing cognitively, socially, and emotionally. Prior to discharge home, caregivers are randomly selected to receive either standard care (typical support and/or resources) or standard care plus problem-based telephone counseling.

The telephone follow-up group receives a telephone call from a caregiver support specialist at 2, 4, 6, 8, 10, 12, 14, and 16 weeks after discharge of the patient with TBI home with the option of two additional calls. During those calls, the caregiver support specialist provides training on problem-solving skills along with education on topics of interest to caregivers of persons with TBI.

An outcome assessment is done at 6 months and 1 year after discharge home.

ELIGIBILITY:
Inclusion Criteria:

* Family member or other person having a long-term relationship (at least one year) with person with TBI admitted to hospital and discharged home from acute care, inpatient rehabilitation, and/or skilled nursing facility within 7 months of date of injury.
* Sufficient English to permit communication without an interpreter.

Exclusion Criteria:

* Lack of a telephone.
* Lack of a permanent home address.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-06; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Composite measure based on the Bakas Caregiving Outcomes Scale and the Brief Symptom Inventory | 6 mos and 1 year post discharge home

SECONDARY OUTCOMES:
Caregiver community participation as measured by the PART-O | 6 mos and 1 year post discharge home
Caregiver employment | 6 mos and 1 year post discharge home
Caregiver resource utilization | 6 mos and 1 year post discharge home
Perceived Quality of Life (person with TBI) | 6 mos post discharge home
Brief Symptom Inventory (person with TBI) | 6 mos post discharge home

CONTACTS AND LOCATIONS:
Overall Officials: Janet M. Powell, PhD, Principal Investigator — University of Washington; Kathleen R. Bell, MD, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Powell JM, Wise EK, Brockway JA, Fraser R, Temkin N, Bell KR. Characteristics and Concerns of Caregivers of Adults With Traumatic Brain Injury. J Head Trauma Rehabil. 2017 Jan/Feb;32(1):E33-E41. doi: 10.1097/HTR.0000000000000219. PMID 27022956
- [Derived] Powell JM, Fraser R, Brockway JA, Temkin N, Bell KR. A Telehealth Approach to Caregiver Self-Management Following Traumatic Brain Injury: A Randomized Controlled Trial. J Head Trauma Rehabil. 2016 May-Jun;31(3):180-90. doi: 10.1097/HTR.0000000000000167. PMID 26394294